CLINICAL TRIAL: NCT06131281
Title: Comparing Outcomes of Classic Transoral Outlet Reduction (TORe) Versus Endoscopic Submucosal Dissection-TORe: A Randomized Controlled Trial
Brief Title: Comparing Reduction With ESD- Versus APC-TORe
Acronym: CREATORe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stephen Firkins (Other)
Responsible Party: Sponsor-Investigator, Stephen Firkins, Co-Director of Bariatric Endoscopy, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-886
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Roux-en-y Anastomosis Site; Weight Gain
MeSH Terms: conditions — Obesity; Weight Gain

STUDY DESIGN:
Intervention Model Description: Prospective, single-blinded, randomized controlled trial
Who Masked: Participant
Masking Description: Participants will be blinded to which procedure they received. The physician performing the procedure cannot be blinded to the procedure type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- E-TORe (Experimental): Participants in this arm received the E-TORe procedure
  Interventions: Procedure: E-TORe
- c-TORe (Active Comparator): Participants in this arm received the "classical" or c-TORe procedure
  Interventions: Procedure: c-TORe

INTERVENTIONS:
Procedure: E-TORe — The E-TORe utilizes ESD in addition to APC prior to endoscopic suturing. In this approach, a standardized solution of normal saline or hetastarch mixed with methylene blue and epinephrine is injected into the gastric rim of the GJA outlet. The mucosa is then carefully incised to expose the underlying muscular layer for a width of approximately 1cm around the GJA circumference. Following ESD, APC is then applied to the inner and outer mucosal margins of the ESD tract. Finally, endoscopic sutures are then placed in purse string fashion and cinched closed around a 6mm TTS balloon.
  Other Names: ESD-TORe, endoscopic submucosal dissection TORe
  Arms: E-TORe
Procedure: c-TORe — The c-TORe will be completed utilizing APC prior to endoscopic suturing. In this approach, the gastric rim of the anastomosis is circumferentially ablated using APC (forced APC, flow of 0.8 L/min and power of 30-70 watts) extending an average of 1-2 cm from the outlet. Following ablation, endoscopic sutures are placed in a purse string fashion within the ablated area and the outlet cinched closed over a 6mm through-the scope (TTS) balloon.
  Other Names: classic TORe, APC-TORe, argon plasma coagulation TORe
  Arms: c-TORe

SUMMARY:
The goal of this clinical trial is to compare two variations of the same procedure used to assist with weight loss in patients who have a history of Roux-en-Y gastric bypass who have experienced weight regain. The procedure being studied is called the Transoral Outlet Reduction (TORe), and the trial will compare two different ways to complete the TORe procedure. The main question[s] it aims to answer are:

* Which variation of the TORe procedure results in more weight loss?
* Which variation of the TORe is safer? Participants who are eligible and willing to undergo the TORe procedure to assist with weight loss will have the procedure completed either one of the two ways. All other care will be exactly the same between the two groups. Researchers will compare outcomes between the two procedure variations, looking at which one results in more weight loss, is more successful, and safer.

DETAILED DESCRIPTION:
Weight regain after having a Roux-en-Y gastric bypass is common. One of the primary reasons for weight regain after bypass is stretching out or "dilation" of the surgical connection created between what is left of the stomach and the small intestine (called the anastamosis). As the ability to suture with the help of a scope inserted through the mouth into the stomach instead of surgery, the transoral outlet reduction (TORe) was developed. The TORe involves suturing around the stretched out anastamosis, allowing it to be pulled tighter and shrink down, resulting in weight loss, and is an entirely endoscopic and reversible procedure. As the procedure advanced, "burning" of the stomach lining using a technique called argon plasma coagulation (APC), in addition to suturing, became the standard way to perform the TORe procedure. The APC helps the stomach tissue shrink even more and heal into place better, causing even more weight loss. This is now the classic way to perform the TORe (hereby called the "c-TORe"), and is now widely used to help patients who have regained weight after gastric bypass.

Multiple studies report the c-TORe results in an average of 8-9% total body weight loss. However more recently, another variation of the TORe was developed, which uses endoscopic submucosal dissection (ESD). In the ESD-TORe (hereby called the E-TORe), the physician makes a small cut in the surface layer of the anastamosis in addition to APC and suturing. In the only study comparing c-TORe to E-TORe, E-TORe resulted in significantly more weight loss. However, there are several limitations to this study that require more investigation.

This clinical trial will compare the c-TORe and the E-TORe. Patients who are eligible and willing to undergo a TORe procedure will be assigned to get either the c-TORe or the E-TORe. They will undergo the procedure with a physician experienced in both types of the procedure. Participants will be followed for one year after the procedure to compare which procedure type results in more weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with history of Roux-en-Y gastric bypass and weight regain
* Dilated gastrojejunal anastamosis as diagnosed on endoscopy
* Patients undergoing standard of care for treatment of obesity with endoscopic revisional procedure (a.k.a. TORe) who are enrolled in the GI Bariatric Endoscopy program and clinic at the study site

Exclusion Criteria:

* Prior revision of gastric bypass
* Active and uncontrolled gastro-esophageal reflux disease defined as ≥ grade C esophagitis
* Active untreated Helicobacter pylori infection
* Malignancy newly diagnosed by endoscopy
* Upper gastro-intestinal conditions such as ulcers, polyps, gastric varices, strictures, congenital or acquired intestinal telangiectasia or other abnormalities that preclude completion of TORe
* Presence of gastrogastric or gastroenteric fistula
* Inability to undergo general anesthesia
* Participating in another ongoing clinical trial of an investigational weight loss drug or device
* Active pregnancy
* Use of anticoagulation therapy or P2Y12 inhibitors which cannot be discontinued for the time frame surrounding the procedure
* Insulin-dependent diabetes mellitus
* Unwillingness to comply with standard post-TORe dietary guidelines and follow-up care
* Any other anatomical, technical or otherwise factor that limits the ability of the endoscopist to perform either E-TORe or c-TORe
* Any additional factor, which in the investigator's opinion, might jeopardize the subject's safety or compliance with the trial protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Weight change at 6 months | 6 months from procedure date
  Percent total body weight change 6 months following TORe procedure
Weight change at 12 months | 12 months from procedure date
  Percent total body weight change 12 months following TORe procedure

SECONDARY OUTCOMES:
Technical success | Day of procedure
  Rates of technical success of the procedure as determined by the experienced endoscopist performing the TORe procedure
Procedure time | Day of procedure
  Mean time to complete each procedure type
Adverse event rate | One year from date of procedure
  Rate of adverse events related to each procedure type
5% total body weight loss | One year from date of procedure
  Proportion of subjects who achieved at least 5% total body weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Firkins, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clapp B, Ponce J, DeMaria E, Ghanem O, Hutter M, Kothari S, LaMasters T, Kurian M, English W. American Society for Metabolic and Bariatric Surgery 2020 estimate of metabolic and bariatric procedures performed in the United States. Surg Obes Relat Dis. 2022 Sep;18(9):1134-1140. doi: 10.1016/j.soard.2022.06.284. Epub 2022 Jun 26. PMID 35970741
- [Background] Karmali S, Brar B, Shi X, Sharma AM, de Gara C, Birch DW. Weight recidivism post-bariatric surgery: a systematic review. Obes Surg. 2013 Nov;23(11):1922-33. doi: 10.1007/s11695-013-1070-4. PMID 23996349
- [Background] El Ansari W, Elhag W. Weight Regain and Insufficient Weight Loss After Bariatric Surgery: Definitions, Prevalence, Mechanisms, Predictors, Prevention and Management Strategies, and Knowledge Gaps-a Scoping Review. Obes Surg. 2021 Apr;31(4):1755-1766. doi: 10.1007/s11695-020-05160-5. Epub 2021 Feb 8. PMID 33555451
- [Background] Athanasiadis DI, Martin A, Kapsampelis P, Monfared S, Stefanidis D. Factors associated with weight regain post-bariatric surgery: a systematic review. Surg Endosc. 2021 Aug;35(8):4069-4084. doi: 10.1007/s00464-021-08329-w. Epub 2021 Mar 1. PMID 33650001
- [Background] Bastos EC, Barbosa EM, Soriano GM, dos Santos EA, Vasconcelos SM. Determinants of weight regain after bariatric surgery. Arq Bras Cir Dig. 2013;26 Suppl 1:26-32. doi: 10.1590/s0102-67202013000600007. English, Portuguese. PMID 24463895
- [Background] Runge TM, Jirapinyo P, Chan WW, Thompson CC. Dysphagia predicts greater weight regain after Roux-en-Y gastric bypass: a longitudinal case-matched study. Surg Obes Relat Dis. 2019 Dec;15(12):2045-2051. doi: 10.1016/j.soard.2019.06.041. Epub 2019 Jul 9. PMID 31931976
- [Background] Abu Dayyeh BK, Lautz DB, Thompson CC. Gastrojejunal stoma diameter predicts weight regain after Roux-en-Y gastric bypass. Clin Gastroenterol Hepatol. 2011 Mar;9(3):228-33. doi: 10.1016/j.cgh.2010.11.004. Epub 2010 Nov 17. PMID 21092760
- [Background] Jense MTF, Palm-Meinders IH, Sigterman-Nelissen R, Boerma EG, Liem RSL, Swank DJ, Greve JWM. The Benefits of Banded over Non-banded Roux-en-Y Gastric Bypass in Patients with Morbid Obesity: a Multi-center Study. Obes Surg. 2022 Jun;32(6):1856-1863. doi: 10.1007/s11695-022-06024-w. Epub 2022 Apr 2. PMID 35366739
- [Background] Thompson CC, Chand B, Chen YK, DeMarco DC, Miller L, Schweitzer M, Rothstein RI, Lautz DB, Slattery J, Ryan MB, Brethauer S, Schauer P, Mitchell MC, Starpoli A, Haber GB, Catalano MF, Edmundowicz S, Fagnant AM, Kaplan LM, Roslin MS. Endoscopic suturing for transoral outlet reduction increases weight loss after Roux-en-Y gastric bypass surgery. Gastroenterology. 2013 Jul;145(1):129-137.e3. doi: 10.1053/j.gastro.2013.04.002. Epub 2013 Apr 5. PMID 23567348
- [Background] Jirapinyo P, Kumar N, AlSamman MA, Thompson CC. Five-year outcomes of transoral outlet reduction for the treatment of weight regain after Roux-en-Y gastric bypass. Gastrointest Endosc. 2020 May;91(5):1067-1073. doi: 10.1016/j.gie.2019.11.044. Epub 2019 Dec 7. PMID 31816315
- [Background] Schulman AR, Kumar N, Thompson CC. Transoral outlet reduction: a comparison of purse-string with interrupted stitch technique. Gastrointest Endosc. 2018 May;87(5):1222-1228. doi: 10.1016/j.gie.2017.10.034. Epub 2017 Nov 3. PMID 29108984
- [Background] Dhindsa BS, Saghir SM, Naga Y, Dhaliwal A, Ramai D, Cross C, Singh S, Bhat I, Adler DG. Efficacy of transoral outlet reduction in Roux-en-Y gastric bypass patients to promote weight loss: a systematic review and meta-analysis. Endosc Int Open. 2020 Oct;8(10):E1332-E1340. doi: 10.1055/a-1214-5822. Epub 2020 Sep 22. PMID 33015335
- [Background] Jirapinyo P, de Moura DTH, Thompson CC. Endoscopic submucosal dissection with suturing for the treatment of weight regain after gastric bypass: outcomes and comparison with traditional transoral outlet reduction (with video). Gastrointest Endosc. 2020 Jun;91(6):1282-1288. doi: 10.1016/j.gie.2020.01.036. Epub 2020 Jan 31. PMID 32007520
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/81/NCT06131281/Prot_SAP_000.pdf